CLINICAL TRIAL: NCT00051103
Title: An Open-Label, Multicenter, Single Arm Phase II Study of Oral GW572016 as Single Agent Therapy in Subjects With Advanced or Metastatic Breast Cancer Who Have Progressed While Receiving Herceptin Containing Regimens
Brief Title: Oral Drug Study In Women With Refractory Metastatic Breast Cancer After First-line or Second-line Herceptin.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF 20002; NCT00044330 (obsolete NCT alias); NCT00053066 (obsolete NCT alias)
Record Dates: First submitted 2003-01-03; First posted 2003-01-06 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Breast Cancer; Neoplasms, Breast
Keywords: Refractory
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: Investigational Cancer Drug

SUMMARY:
The purpose of this study is to determine the efficacy of an oral investigational drug for the treatment of metastatic breast cancer tumors that are known to overexpress HER2/neu.

ELIGIBILITY:
Inclusion Criteria: (The patient must meet the following criteria in order to be eligible for this study.)

* Signed informed consent
* No more than two prior regimens for metastatic breast cancer. Each regimen must have contained Herceptin.
* Refractory Stage IIIb or IV breast cancer
* HER2/neu tumor overexpression
* Disease progression while receiving a prior chemotherapy regimen with Herceptin alone or in combination with other chemotherapy.
* Tumor tissue available for testing.
* 2 weeks since treatment with Herceptin (alone or in combination).
* Able to swallow and retain oral medication
* Cardiac ejection fraction within the institutional range of normal as measured by MUGA (Multiple Gated Acquisition Scan).
* Adequate kidney and liver function
* Adequate bone marrow function

Exclusion Criteria: (The patient cannot meet any of the following criteria in order to be eligible for this study.)

* Prior regimens did not include Herceptin.
* Pregnant or lactating.
* Conditions that would affect absorption of an oral drug
* Serious medical or psychiatric disorder that would interfere with the patient's safety or informed consent.
* Severe cardiovascular disease or cardiac disease requiring a device.
* Active infection.
* Brain metastases.
* Concurrent cancer therapy or investigational therapy.
* Use of oral or IV steroids.
* Unresolved or unstable serious toxicity from prior therapy.
* Treatment with EGFR (Endothelial Growth Factor Receptor) inhibitor other than Herceptin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (27):
- United States (27):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Bettendorf, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Hooksett, New Hampshire
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salem, Virginia

REFERENCES:
- [Background] Blackwell KL, Pegram MD, Tan-Chiu E, Schwartzberg LS, Arbushites MC, Maltzman JD, Forster JK, Rubin SD, Stein SH, Burstein HJ. Single-agent lapatinib for HER2-overexpressing advanced or metastatic breast cancer that progressed on first- or second-line trastuzumab-containing regimens. Ann Oncol. 2009 Jun;20(6):1026-31. doi: 10.1093/annonc/mdn759. Epub 2009 Jan 29. PMID 19179558
- See also: A website where viewers can complete a clinical study-matching questionnaire and also sign up for future study notification and healthcare newsletters. — http://www.findclinicalstudy.com/rdt.cfm?R=gov&d=642&t=1